CLINICAL TRIAL: NCT01881503
Title: Expanded Access Protocol for the Treatment Use of HBOC-201
Brief Title: Expanded Access Study of HBOC-201 (Hemopure) for the Treatment of Life-Threatening Anemia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Collaborators: HbO2 Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-12-454
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2021-08

CONDITIONS: Anemia
Keywords: life-threatening anemia; blood alternative; HBOC
MeSH Terms: conditions — Anemia | interventions — HBOC 201

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Other): all qualifying subjects will receive HBOC-201 (Hemopure) to treat their life-threatening anemia
  Interventions: Biological: HBOC-201

INTERVENTIONS:
Biological: HBOC-201 — HBOC-201 is purified, cross-linked, acellular bovine hemoglobin (Hb) in a modified lactated Ringer's solution.
  Other Names: Hemopure

SUMMARY:
The purpose of this expanded access study is to be able to provide treatment with HBOC-201 to patients with life-threatening anemia for whom blood is not an option.

HBOC-201 is not FDA approved for use in the United States, but is approved as an oxygen carrier in South Africa and Russia.

DETAILED DESCRIPTION:
i. Initial Dose

For patients with a hemoglobin level less than 6 mg/dl, an initial dose of 32.5 g (one unit) of HBOC 201 is recommended, to be followed by infusion of additional units as necessary to achieve and maintain a total hemoglobin concentration above 6 g/dl, provided that the patient's circulatory volume is properly controlled and will not impose an inappropriate risk.

ii. Subsequent Doses

The need for additional dose administration should be assessed after each infusion as clinically indicated.

Dosing will be stopped if any one of the following occurs:

* resolution of critical ischemia
* death
* recovery of native Hemoglobin levels to > 6 g/dL,
* evidence of reticulocytosis

ELIGIBILITY:
Inclusion Criteria:

1. Patients > = 18 years of age
2. Patients with hemoglobin < = 8g/dL with with active bleeding, physiologic evidence of critical ischemia, for example: elevated troponins, altered mental status, acute renal failure, lactic acidosis or central nervous system supply dependency
3. Patients or their Legally Authorized Representatives who are able and willing to provide informed consent

Exclusion Criteria:

1. Patients with known hypersensitivity or allergy to beef products
2. Patients with pre-existing uncontrolled hypertension, heart failure, renal failure, circulatory hypervolemia or systemic mastocytosis (on a case by case and quality of life determination)
3. Patients > 80 years of age (on a case by case and quality of life determination)
4. Patients who are eligible for blood transfusions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
survival | 1 week
  subjects will receive HBOC-201 to treat life-threatening anemia

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Gianatiempo, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.englewoodhealth.org